CLINICAL TRIAL: NCT06035185
Title: The Effect of Apical Enlargement on Microbial Load Before and After Passive Ultrasonic Activation in Asymptomatic Teeth Periapical Lesions
Brief Title: Microbial Load After Apical Enlargement in Asymptomatic Teeth With Periapical Lesion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Tan Firat Eyuboglu, Associate Professor, Istanbul Medipol University Hospital
Other Study IDs: IMU-2023
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Root Canal Infection; Periapical Diseases; Periapical; Infection; Endodontic Disease
Keywords: apical shaping; Droplet Digital PCR; irrigation activation; microbial load; root canal cleanliness
MeSH Terms: conditions — Periapical Diseases; Infections; Dental Pulp Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1- One Curve Mini 25/0.4: Root canal shaping will be completed with a heat-treated nickel titanium OneCurve Mini #25/0.4 rotary file (Micro-Mega, Besancon, France) after reaching the apical region with #10 K stainless steel files (Dentsply Maillefer, Ballaigues, Switzerland). The irrigation solution will be used by adapting an ultrasonic tip (IRRI S 21/25; VDW, Munich, Germany) to an ultrasonic device (VDW Ultra; VDW, Munich, Germany). The tip will be activated a total of three times, each cycle lasting 20 s and involving the use of 1 ml of 3% NaOCl. Then 2 ml of 17% EDTA solution will be activated for 1 minute as described above. The ultrasonic tip will be placed 2 mm shorter than the working length without touching the canal walls.
  Interventions: Procedure: apical shaping size
- Group 2- One Curve Mini 35/0.4: Root canal shaping will be completed with a heat-treated nickel titanium OneCurve Mini #35/0.4 rotary file (Micro-Mega, Besancon, France) after reaching the apical region with #10 K stainless steel files (Dentsply Maillefer, Ballaigues, Switzerland). The irrigation solution will be used by adapting an ultrasonic tip (IRRI S 21/25; VDW, Munich, Germany) to an ultrasonic device (VDW Ultra; VDW, Munich, Germany). The tip will be activated a total of three times, each cycle lasting 20 s and involving the use of 1 ml of 3% NaOCl. Then 2 ml of 17% EDTA solution will be activated for 1 minute as described above. The ultrasonic tip will be placed 2 mm shorter than the working length without touching the canal walls.
  Interventions: Procedure: apical shaping size

INTERVENTIONS:
Procedure: apical shaping size — 24 patients will randomly be assigned to two groups according to the apical shaping size during root canal treatment: 25/.04 and 35/.04. Microbiological sampling of the teeth will be done with paper cones in three steps during the root canal treatment: 1. Sterility control samples (SR1) from the tooth surface after cavity preparation, 2. The first microbiological sample (S1) from the root canal after the initial file reaches the working length. 3. The second microbiological sample (S2) from the root canal after the shaping and irrigation of the root canal is finished. 4. The third microbiological sample (S3) from the root canal after the irrigation activation in the root canal is finished.The samples will be sent to the genetic analysis laboratory for further analysis in the cold chain using a Droplet Digital PCR.

SUMMARY:
The goal of this observational study is to define the role of apical shaping and irrigation activation on root canal cleanliness. The main questions it aims to answer are:

* does the effectiveness of irrigation activation depends on apical shaping?
* can a similar success be achieved by increasing apical shaping without irrigation activation Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items].

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of apical enlargement with two different diameters on the intraradicular microbiota of teeth with chronic apical periodontitis lesion before and after passive ultrasonic irrigation activation using ddPCR analysis in vivo.The study was planned as a randomized controlled clinical trial. We are planning to include 24 patients who was referred to the Istanbul Medipol University Faculty of Dentistry Endodontic Clinic with the need for root canal treatment, with asymptomatic chronic apical periodontitis. 24 patients will randomly be assigned to two groups according to the apical shaping size during root canal treatment: 25/.04 and 35/.04. Microbiological sampling of the teeth will be done with paper cones in three steps during the root canal treatment: 1. Sterility control samples (SR1) from the tooth surface after cavity preparation, 2. The first microbiological sample (S1) from the root canal after the initial file reaches the working length. 3. The second microbiological sample (S2) from the root canal after the shaping and irrigation of the root canal is finished. 4. The third microbiological sample (S3) from the root canal after the irrigation activation in the root canal is finished.The samples will be sent to the genetic analysis laboratory for further analysis in the cold chain using a Droplet Digital PCR.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65
* Patients complying with the ASA1 and ASA2 classification (American Society of Anesthesiology)
* Patients who has molar teeth with radiolucent lesions in the periapical region
* The volunteer himself/herself or his/her legal representative wants to participate in the research by signing the 'Voluntary Consent Form'.
* Being able to tolerate the treatment physically and mentally

Exclusion Criteria:

* Patients who have taken antibiotics/corticosteroids in the last 3 months
* Patients with systemic disease
* Teeth that cannot be properly isolated with a rubber dam
* Teeth without coronal sealing,
* Teeth with periodontal pocket depth>4 mm and teeth with crown / root fracture.
* Individuals who continue or are considering starting orthodontic treatment during the research
* Pregnant and lactating individuals
* The volunteer himself/herself or his/her legal representative does not want to participate in the research by signing the 'Voluntary Consent Form'.
* Teeth that are damaged enough to require post-core treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 24 patients who was referred to the Istanbul Medipol University Faculty of Dentistry Endodontic Clinic with the need for root canal treatment, with asymptomatic chronic apical periodontitis, witj clinical and radiographic findings. The study will be carried out in Istanbul Medipol University Faculty of Dentistry Endodontic Clinic, and patients with appropriate criteria will be informed about the treatment to be performed and their consent will be obtained. In this observational type study, patients treated by the same physician will be followed.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
apical shaping size | through study completion, an average of 1 year
  does apical shaping size affect the microbial load in the root canal after shaping and irrigation finishes? microbial load after two different apical shaping size will be compared between two groups. Droplet Digital PCR will be used to measure and compare the microbial load within the root canal before and after irrigation protocol in each group to measure this outcome.
irrigation activation | through study completion, an average of 1 year
  does irrigation activation affect the microbial load in the root canal? microbial load after chemomechanical cleaning of the root canal and after the irrigation activation will be compared. Droplet Digital PCR will be used to measure microbial load before after irrigation activation in each canal to see its effect on reduction fo microbial load within the root canal.

SECONDARY OUTCOMES:
the effect of apical shaping in irrigation activation | through study completion, an average of 1 year
  does apical size affect the irrigation activation? the microbial load after chemomechanical cleaning of the root canal and after irrigation activation will be compared between two groups (with different apical shaping size) to analyse the effect of apical shaping on irrigation activation. Droplet Digital PCR results before and after irrigation activation in root canals with different apical size will be compared to measure this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tan Firat Eyüboglu, PhD, JSD, Principal Investigator — Istanbul Medipol University Hospital
Locations (1):
- Istanbul Medipol University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
due to regulatory reasons the participant data will not be shared.